CLINICAL TRIAL: NCT05656482
Title: Evaluation of the Ability of a Cat Food to Reduce Respiratory Symptoms in Cat Allergic Patients: Pilot Study
Brief Title: Ability of a Cat Food to Reduce Respiratory Symptoms in Cat Allergic Patients
Acronym: CATS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MASK-air SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: KM00232
Record Dates: First submitted 2022-12-05; First posted 2022-12-19 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cats fed with PRO PLAN® LIVECLEAT® — Patient with domestic cats fed with an egg product containing anti-Fel d1 IgY (PRO PLAN® LIVECLEAT®)

SUMMARY:
Cat allergy is the most common animal allergy, affecting approximately 1 in 5 adults worldwide. The prevalence of allergy to furry animals is increasing, and cat allergy is a major risk factor for the development of asthma and rhinitis.

Fel-d1 is the major feline allergen, to which 95% of cat allergic people react. All cats produce Fel-d1 regardless of breed, age, coat type, sex or weight. Fel-d1 is contained primarily in the saliva and sebum of cats.

This allergy manifests itself as allergic rhinitis (AR) (sneezing, cold, coughing, conjunctivitis with watering and itching), severe asthma, and irritation and swelling of the skin when scratched.

A new approach to managing cat allergies is to neutralize the allergens at the source by feeding domestic cats a diet containing anti-Fel-d1 IgY antibodies. The purpose of this pilot study is to determine whether feeding domestic cats a food containing an egg product with anti-Fel d1 IgY (PRO PLAN® LIVECLEAT®) induces a reduction of allergic symptoms in their owners.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled allergic rhinitis (with or without treatment)
* Persistent allergic rhinitis with worsening of symptoms upon exposure to cats
* Presence of one or two cats in the household, whose diet consists mainly of dry kibble
* Agreement of the patient to change the food of the cat(s) and to feed it exclusively with the test kibbles during the study.
* Diagnosis of cat allergy defined by a positive prick test to standardized cat allergen or cat-specific IgE.
* Absence of allergy to pollens emitted in the region during the 4 months following the inclusion date, confirmed by a negative skin test.
* Person owning an android and/or IOS smartphone and having the possibility to connect to the internet (via phone subscription or WIFI connection),
* Person who agrees to install the MASK-air application (medical device) on his personal smartphone,
* Person having read and understood the information note and having signed their participation agreement before any specific procedure of the study.

Exclusion Criteria:

* Person planning to be away from the cat(s) for more than one week/month in the 4 months following the inclusion visit
* Patient who has had a new cat in the home for less than one month
* Patient in regular contact with other animals to which they are allergic
* Patient with uncontrolled asthma
* Patient receiving immunotherapy for cat allergies
* Patient participating or having participated in an allergic rhinitis study within the last 30 days or 5 half-lives of study medication
* Person who has difficulty understanding or reading the information
* Person declaring to be under guardianship, curatorship or safeguard of justice.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: a total of 50 Allergic patient to cats is expected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Change of the global Visual Analogic Scale (VAS) mean from Baseline period (Day 0- Day 15) at end period (Day 98-Day112) | Baseline (Day 0- Day 15) and observation period (Day 98-Day112)
  The approach will be considered beneficial if there is a statistically significant decrease in this criterion on the D98-J112 period compared to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Pham-Thi, Dr, Principal Investigator — Allergologist
Locations (1):
- Cabinet médical Lion de Raspail, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bousquet J, Gherasim A, de Blay F, Mathieu-Dupas E, Batot G, Laune D, Sousa-Pinto B, Zuberbier T, Pham-Thi N; MASK-cat study group. Proof-of-concept study of anti-Fel d 1 IgY antibodies in cat food using the MASK-air(R) app. Clin Transl Allergy. 2024 May;14(5):e12353. doi: 10.1002/clt2.12353. PMID 38676659